CLINICAL TRIAL: NCT05839431
Title: Virtual Reality for Youth Phobias
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: The Children's Trust, Miami FL (Other)
Responsible Party: Principal Investigator, Jill May Ehrenreich, Professor, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20221240
Record Dates: First submitted 2023-04-20; First posted 2023-05-03 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Specific Phobia; Social Anxiety Disorder; Autism Spectrum Disorder
Keywords: Virtual Reality
MeSH Terms: conditions — Phobia, Specific; Phobia, Social; Autism Spectrum Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Therapy for Youth Phobias (Experimental): Participants will undergo up to 10 weeks of virtual reality-assisted exposure therapy.
  Interventions: Behavioral: Virtual Reality for Youth Phobias

INTERVENTIONS:
Behavioral: Virtual Reality for Youth Phobias — The intervention will consist of up to 10, 50-minute-long weekly in-person individual sessions of virtual reality-assisted exposure therapy. This intervention also includes psychoeducation about anxiety/phobias and their maintenance, youth strategies for tolerating distress, and parent strategies for reducing accommodation of anxiety.

SUMMARY:
The purpose of this study is to examine the effectiveness of virtual reality (VR) delivered exposure therapy for youth with phobias or social anxiety, with and without autism spectrum disorder. The study team is also interested in collecting information to better understand phobias and social anxiety.

ELIGIBILITY:
Inclusion Criteria:

1. The target population for this project are 48 youth (ages of 8-16) that meet criteria for a specific phobia or social anxiety disorder within Miami-Dade County.
2. Youth will be eligible if they or their parent report clinically significant symptoms of social anxiety disorder or a specific phobia targeted with the VR program, based on self- or parent-report scores on online screening measures (>1 average total scores on Severity Measure for Specific Phobia-Child or Social Anxiety Disorder-Child) or clinician-report diagnosis (i.e., diagnosed with Social Anxiety Disorder or Specific Phobia during clinical interview).
3. Youth are able to complete study procedures, speak/read English or Spanish sufficiently.
4. Youth have at least one caregiver who can complete all study measures in English or Spanish.
5. Youth have a caregiver who is available to sign study consent forms, remain present during assessments, and fill out study questionnaires.

Exclusion Criteria:

1. Youth who would be inappropriate for a brief VR-exposure therapy protocol will be referred to local resources for additional support or provided with alternate cognitive behavioral therapy services through the clinical center in which this program takes place.
2. Research staff will review all measures and the youth's psychological history and consult with the PI to ensure that the participant does not have a current diagnosis of psychosis, bipolar disorder, acute suicidality, alcohol/substance dependence, or eating disorder.
3. Youth will also be excluded if they are currently receiving psychotherapy elsewhere.
4. Youth with co-occurring intellectual disability may be eligible, but youth who are non-verbal will not be eligible, as some verbal abilities are necessary in order to communicate with the clinician during the intervention.
5. Youth who are currently suicidal or who have engaged in suicidal behaviors within the past 6 months will be excluded (or discussed on a case-by-case basis).
6. Youth who engage in self-harm behaviors (e.g., cutting) and who do not present with suicidal intent will be allowed to participate.
7. If youth develop psychiatric problems (e.g., severe depression, acute suicidal ideation/intent, severe conduct problems) that require a higher level of care, youth will be withdrawn from the study and referred for appropriate treatment.
8. Youth currently taking psychotropic medication for a co-morbid psychiatric illness will be included without a wash-out period (to not delay intervention).

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire | Up to 10 weeks
  The Client Satisfaction Questionnaire is an 8-item measure of client satisfaction with services with both a parent and child version. The total scores range from 8 to 32, with higher scores indicating higher satisfaction.

SECONDARY OUTCOMES:
Change in social anxiety as measured by the Severity Measure for Social Anxiety Disorder (Social Phobia) | Baseline, 10 weeks
  The Severity Measure for Social Anxiety Disorder (Social Phobia)-Child is a 10-item measure that assesses the severity of symptoms of social anxiety (social phobia) in children and adolescents over the last 7 days. Scores range from 0 to 4. An average total score of 2 or greater indicates at least moderate social anxiety.
Change in social anxiety as measured by the Severity Measure for Specific Phobia | Baseline, 10 weeks
  The Severity Measure for Specific Phobia-Child is a 10-item measure that assesses the severity of symptoms of specific phobias in children and adolescents, including those targeted by the VR programs, over the last 7 days. Scores range from 0 to 4. An average total score of 2 or greater indicates at least moderate phobia symptoms.
Change in intolerance of uncertainty as measured by the Intolerance of Uncertainty Scale for Children | Baseline, 10 weeks
  The Intolerance of Uncertainty Scale for Children 12-item child and parent report of the tendency to react negatively on an emotional, cognitive, and/or behavioral level to uncertain situations and events. Scores range from 12 to 60. Higher scores indicate greater intolerance of uncertainty.
Change in family accommodation as measured by the Family Accommodation Scale-Anxiety | Baseline, 10 weeks
  The Family Accommodation Scale-Anxiety is a 9-item scale of measuring caregiver accommodation behaviors (modification of routines, facilitating avoidance, etc.) in light of youth anxiety. Scores range from 0 to 36. Higher scores indicate greater family accommodation.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Ehrenreich-May, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Coral Gables, Florida, United States

IPD SHARING:
Plan to Share IPD: No